CLINICAL TRIAL: NCT02606838
Title: User Performance of the Styx Lancing System
Brief Title: Evaluation of an Ascensia Lancing System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GCA-2014-001-01
Record Dates: First submitted 2015-11-13; First posted 2015-11-17 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2016-12

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Persons with Diabetes (Experimental): Untrained Persons with Diabetes used the Styx Lancing Device System to obtain fingerstick and Alternate Site palm capillary blood.
  Interventions: Device: Styx Lancing Device

INTERVENTIONS:
Device: Styx Lancing Device — Untrained Persons With Diabetes used the Styx Lancing Device with 28 and 30 Gauge lancets to obtain fingerstick and Alternate Site palm capillary blood. Study Staff tested the capillary blood using Contour NEXT Blood Glucose Meters (BGMs) and recorded the results. Meter results could be numeric, non-numeric (ie, error messages), or not obtained at all.

SUMMARY:
The purpose of this study was to determine if untrained subjects with diabetes could perform basic tasks with the Styx lancing device to obtain adequate blood volume from fingerstick and palm lancings for Blood Glucose Meter testing.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years of age and older
* People with type 1 or type 2 diabetes
* People who regularly perform self-tests (at least once/day) with their own lancing device
* Able to speak, read, and understand English
* Willing to complete all study procedures

Exclusion Criteria:

* Those with missing tips of the fingers indicated in the protocol or physically unable to lance the palm areas and all the fingers indicated in the protocol.
* Hemophilia or any other bleeding disorder
* Pregnancy
* Physical, visual or neurological impairments that would make the person unable to perform testing
* Persons who have used the Styx device in a previous clinical evaluation
* Working for a competitive medical device company, or having an immediate family member who works for such a company
* A condition which, in the opinion of the investigator or designee, would put the person or study conduct at risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Morin, MD, Principal Investigator — Ascensia Diabetes Care
Locations (1):
- Ascensia Diabetes Care, Mishawaka, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Persons With Diabetes
Started | 119
Completed | 119
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Persons With Diabetes
Number analyzed (Participants) | 119
Age, Continuous [Mean (Full Range); unit: years] | 55.1 [23 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 110
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 97
  More than one race | 1
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 119

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Numeric Meter Results When Users Obtain Fingerstick Capillary Blood Using the Styx Lancing Device ( 28 Gauge Lancets)
Description: Untrained subjects with Diabetes operated the Styx Lancing Device with 28 Gauge lancets to obtain fingerstick capillary blood. Study Staff tested the capillary blood using Contour NEXT Blood Glucose Meters (BGMs) and recorded the results. Meter results could be numeric, non-numeric (ie, error messages), or not obtained at all. The number of subjects with numeric BGMS results was determined.
Time Frame: 1 hour
Measure: Number; unit: participants
Groups:
- Persons With Diabetes: Untrained subjects with Diabetes operated the Styx Lancing Device with 28 Gauge lancets to obtain fingerstick capillary blood. Study staff tested the capillary blood using Contour NEXT Blood Glucose Meters (BGMs) and recorded the results. Meter results could be numeric, non-numeric (i.e., error messages), or not obtained at all.
Arm/Group | Persons With Diabetes
Number analyzed (Participants) | 119
participants | 119

2. Secondary Outcome: Number of Subjects With Numeric Meter Results When Users Obtain Alternate Site (AST) Palm Blood Using the Styx Lancing Device ( 28 Gauge Lancets)
Description: Untrained subjects with Diabetes operated the Styx Lancing Device with 28 Gauge lancets to obtain AST palm capillary blood. Study Staff tested the capillary blood using Contour NEXT Blood Glucose Meters (BGMs) and recorded the results. Meter results could be numeric, non-numeric (ie, error messages), or not obtained at all. The number of subjects with numeric BGMS results was determined.
Time Frame: 1 hour
Population: 118 (119-1) Subject results were analyzed. One subject result was not evaluable because staff deviated from protocol by interfering with subject operation of the device.
Measure: Number; unit: participants
Groups:
- Persons With Diabetes: Untrained subjects with Diabetes operated the Styx Lancing Device with 28 Gauge lancets to obtain AST palm capillary blood. Study staff tested the capillary blood using Contour NEXT Blood Glucose Meters (BGMs) and recorded the results. Meter results could be numeric, non-numeric (i.e., error messages), or not obtained at all.
Arm/Group | Persons With Diabetes
Number analyzed (Participants) | 118
participants | 116

3. Secondary Outcome: Number of Subjects With Numeric Meter Results When Users Obtain Fingerstick Capillary Blood Using the Styx Lancing Device ( 30 Gauge Lancets)
Description: Untrained subjects with Diabetes operated the Styx Lancing Device with 30 Gauge lancets to obtain fingerstick capillary blood. Study Staff tested the capillary blood using Contour NEXT Blood Glucose Meters (BGMs) and recorded the results. Meter results could be numeric, non-numeric (ie, error messages), or not obtained at all. The number of subjects with numeric BGMS results was determined.
Time Frame: 1 hour
Measure: Number; unit: participants
Groups:
- Persons With Diabetes: Untrained subjects with Diabetes operated the Styx Lancing Device with 30 Gauge lancets to obtain fingerstick capillary blood. Study staff tested the capillary blood using Contour NEXT Blood Glucose Meters (BGMs) and recorded the results. Meter results could be numeric, non-numeric (i.e., error messages), or not obtained at all.
Arm/Group | Persons With Diabetes
Number analyzed (Participants) | 119
participants | 119

4. Secondary Outcome: Number of Subjects With Numeric Meter Results When Users Obtain Alternate Site (AST) Palm Blood Using the Styx Lancing Device ( 30 Gauge Lancets)
Description: Untrained subjects with Diabetes operated the Styx Lancing Device with 30 Gauge lancets to obtain AST palm capillary blood. Study Staff tested the capillary blood using Contour NEXT Blood Glucose Meters (BGMs) and recorded the results. Meter results could be numeric, non-numeric (ie, error messages), or not obtained at all. The number of subjects with numeric BGMS results was determined.
Time Frame: 1 hour
Population: 117 (119-2) Subject results were analyzed. Two subject results were not evaluable because staff deviated from protocol by interfering with subjects' operation of the device.
Measure: Number; unit: participants
Groups:
- Persons With Diabetes: Untrained subjects with Diabetes operated the Styx Lancing Device with 30 Gauge lancets to obtain AST palm capillary blood. Study staff tested the capillary blood using Contour NEXT Blood Glucose Meters (BGMs) and recorded the results. Meter results could be numeric, non-numeric (i.e., error messages), or not obtained at all.
Arm/Group | Persons With Diabetes
Number analyzed (Participants) | 117
participants | 114

5. Secondary Outcome: Percent of Responses From Persons With Diabetes That Either 'Strongly Agree' or 'Agree' or Are 'Neutral' With Questionnaire Statements Regarding the Styx Lancing Device
Description: Staff obtained responses from persons with Diabetes using short questionnaires to provide feedback on instructions for use and the basic operation of the Styx Lancing Device. Subjects could respond 'Strongly Agree' or 'Agree' or are 'Neutral' or 'Disagree' or 'Strongly Disagree'. The percent of subjects who provided responses that were 'Strongly Agree' or 'Agree' or 'Neutral' about each statement was calculated.
Time Frame: 1 hour
Measure: Number; unit: percentage of participants
Arm/Group | Persons With Diabetes
Number analyzed (Participants) | 119
percentage of participants
  I can follow the device instructional insert | 98.3
  I find the lancing device easy to use | 96.6
  I find it easy to insert the lancet into the devic | 99.2
  I can attach the Black Adjustable Endcap | 100
  I am able to do a fingerstick with this device | 100
  I can remove the Clear AST endcap | 100
  Easy to remove lancet without removing w fingers | 97.5
  I like the overall design of the lancing device | 99.2
  Easy / intuitive to do a fingerstick w this device | 97.5

ADVERSE EVENTS:
Groups:
- Persons With Diabetes: Untrained Persons with Diabetes used the Styx Lancing Device System to obtain fingerstick and Alternate Site palm capillary blood.
  Styx Lancing Device System: Untrained Persons With Diabetes used the Styx Lancing Device with 28 and 30 Gauge lancets to obtain fingerstick and Alternate Site palm capillary blood. Study Staff tested the capillary blood using Contour NEXT Blood Glucose Meters (BGMs) and recorded the results. Meter results could be numeric, non-numeric (ie, error messages), or not obtained at all.
Arm/Group | Persons With Diabetes
Serious Adverse Events (participants affected / at risk) | 0/119
Other Adverse Events (participants affected / at risk) | 1/119
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Persons With Diabetes (N=119)
Hypoglycemia (Endocrine disorders) | 1 (1) — Subject's hypoglycemia was resolved at this visit

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes